CLINICAL TRIAL: NCT03455179
Title: Effects of Slow-speed Traditional Resistance Training, High-speed Resistance Training and Multicomponent Training With Variable Resistances on Molecular, Body Composition, Neuromuscular, Physical Function and Quality of Life Variables in Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Oxidative Pathology Unit of the Department of Biochemistry and Molecular Biology, University of Valencia. (Unknown); City countil of Valencia. Area of Social welfare, Education and Sport, older people section. (Unknown); Municipal Center of Activities for Older People of Campanar, Valencia, Spain (Unknown); Municipal Center of Activities for Older People of Nou Benicalap, Valencia, Spain (Unknown); The Faculty of Nursing and Podiatry, University of Valencia. (Unknown); LabPsiTec (Other); University Clinic of Nutrition, Physical Activity and Physiotherapy CUNAFF, University of Valencia (Unknown); Analclinic: clinical analysis laboratories, Valencia, Spain (Unknown); University Institute of Telematics Medicine, Valencia, Spain (Unknown)
Responsible Party: Principal Investigator, Juan Carlos Colado Sánchez, Full professor of the Department of Physical Education and Sports, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H1508742840440
Record Dates: First submitted 2018-02-21; First posted 2018-03-06 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Aging
Keywords: Older; Physical function; Power training; Oxidative stress; Elastic band; OMNI-RES perceived exertion scale; Strength training

STUDY DESIGN:
Intervention Model Description: This is a randomized, duoble-blind (participant-outcome assessor), 4 arms prospective parrallel desing clinical trial. The older adults will be recruited from the Municipal Activity Centers for Older People located in Valencia and will be randomized in a prospective clinical trial study with a 4 parallel arms study design to a slow-speed traditional resistance training, high-speed resistance training, multicomponent training or control over a 20 weeks period.
Who Masked: Participant, Outcomes Assessor
Masking Description: For masking the participants, the investigators will not inform participants of what group they will be in. For outcome assessor, data collectors and data analysts independent people will be use, and if this is not possible, a random code will be created for each participant so that it is not possible to identify which group belongs to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Slow-speed traditional resistance training (Experimental): Resistance training with variable resistances (elastic band) at high intensity and slow-speed (2s of concentric contraction and 2s of eccentric contraction) twice a week over 20 weeks.
  Interventions: Other: Slow-speed traditional resistance training
- High-speed resistance training (Experimental): Resistance training with variable resistances (elastic band) at low intensity and high-speed (''as fast as possible´´ for the concentric contraction, pause for 1 second and 2-3 seconds for the eccentric contraction) twice a week over 20 weeks.
  Interventions: Other: High-speed resistance training
- Multicomponent training (Experimental): Training sessions with balance, resistance, aerobic, flexibility and coordination components twice a week over 20 weeks.
  Interventions: Other: Multicomponent training
- Control (No Intervention): Participants randomized into the CONTROL group will not undertake any formal intervention and will be asked to maintain their usual physical activity habits and diet.

INTERVENTIONS:
Other: Slow-speed traditional resistance training — The training session will consist in a general warm-up, 6 resistance exercises, including 2 upper limb exercises (elbow curl and chest press), 2 lower limb exercises (lunge and standing hip abduction), and 2 exercises combining both upper and lower limbs at the same time (squat plus upright rowing and squat plus shoulder press) and finally the cooldown routine.The participants will perform in each training session 6 submaximal repetitions equivalent to 85% of the one-repetition maximum (1RM) and 3-4 sets per exercise (high intensity training sessions).
  Arms: Slow-speed traditional resistance training
Other: High-speed resistance training — The participants will perform the same exercises than the TRADICIONAL group with12 submaximal repetitions equivalent to 40-50% 1RM (low-intensity) and 3-4 sets per exercise.
  Other Names: Power training; Explosive resistance training
  Arms: High-speed resistance training
Other: Multicomponent training — Participants will perform, in this order, balance exercises followed by resistance/coordination, aerobic/coordination and flexibility exercises in each session. The balance training will consist in static, dynamic and proactive balance exercises. In the resistance training block, the participants will perform 3-4 sets of 15 submaximal repetitions Participants will perform 2 resistance exercises (squat plus upright rowing and lunge) at traditional slow-speed (2s of concentric contraction and 2s of eccentric contraction).The intensity of the aerobic block will progress from 65 to 85% of the maximum heart rate over the training weeks.
  Arms: Multicomponent training

SUMMARY:
Human aging is characterized by a progressive deterioration of multiple physiologic systems, with marked decreases in skeletal muscle mass, muscle strength, physical function and quality of life beginning in the sixth decade in life. These deleterious modifications have a significant impact upon mobility and ability to undertake daily living activities in elderly people. If we consider that, according to current projections, the proportion of the European population over 65 years will increase from 17% in 2010 to 30% in 2060 and that physical activity participation rates for older adults (>60 years) remain low, with only 16% meeting the recommendations of the American College of Sports Medicine Guidelines (11% for resistance training), we need to understand what type of training (strategy) can be the most effective for reverse physical impairments, and not only that, but which one obtains greater adherence and self-perception for contribute a healthier, active and more independent elderly population in the future.

Thus, the purpose of this study is to investigate the effects of 20-week slow-speed traditional resistance training, high-speed resistance training and multicomponent training program with variable resistance (elastic bands) on molecular, body composition, neuromuscular, physical function and quality of life variables in older adults. This research also aims to evaluate if this novel types of training intervention (using variable resistances such as elastic bands in all the training programs and measure the intensity with the OMNI-RES perceived exertion specific for older adults) is feasible in this population, through analysis of adherence, intervention fidelity and self-perception reported.

DETAILED DESCRIPTION:
Slow-speed traditional resistance training (2-3 seconds for each concentric and eccentric phase) protocols for the elderly have involved relatively heavy loads (70-80% of maximum force) in order to increase strength and function, and has been demonstrated to be an effective strategy to improve biomarkers of health and fitness across a wide range of healthy and clinical older populations, but the results regarding the function are inconsistent in the current literature. However, several studies indicated that muscle power is a stronger predictor than strength for daily motor activities, such as fast walking, stair-climbing, and rising from a chair, and that peak muscle power was associated with functional limitations in older people. Moreover, muscle power declines earlier and at a higher rate than strength. More recently, several authors have designed high-speed resistance training programs, also calling power training or explosive-type resistance training to improve muscle power in older adults rather than strength. However, the effects of high-speed resistance training versus slow-speed traditional resistance training on functional outcomes in older adults are inconsistent, with some studies showing enhanced improvements in function, and others showing no difference in function perhaps because to the application of different training parameters, tests, functional status of the participants or the lengths of the studies. Furthermore, the effects of the high-speed training programs on others variables such as oxidative stress, bone profile or metabolic function are unknown.

On the other hand, current recommendations have recognized that a combination of aerobic activity, strength training and flexibility exercises is important for maintaining physical function in older adults. However, most studies in older individuals have examined the isolated effect of strength and endurance training programs and focused on different health-related fitness parameters. Also, due to the low rates of physical activity in older adults, especially regarding resistance training (11%), it is necessary to study the effects of other types of physical activity possibly more dynamics, like the multicomponent training. Multicomponent training is defined as a well-rounded program that includes endurance, strength, coordination, balance and flexibility exercises and is becoming increasingly popular among the older population and appears to be associated with several health benefits because has the potential to impact both cardiorespiratory and neuromuscular fitness, which both play an important role in maintaining functional fitness and quality of life.

Currently however, there is no evidence which has examined the effectiveness of high-speed resistance training and multicomponent training in older adults (>60 years) in front of slow-speed traditional training not only in respect of the physical function, but also in terms of oxidative stress, bone profile, metabolic status and quality of life. Developing an understanding of novel training strategies can ultimately provide a viable alternative to traditional modes of exercise training for a broader range of participants and increase their adherence to them.

This is a randomized clinical trial (RCT) with 4 parallel arms. The subjects will be divided in 4 groups with a randomized technique: slow-speed traditional resistance training group (TRADITIONAL), high-speed resistance training group (H-SPEED), multicomponent training group (MULTICOMPONENT) and control group (CONTROL). The subjects will be submitted to a 4-session familiarization period and then a 20-week of training program will be performed twice a week.

The TRADITIONAL group will perform 6 submaximal repetitions equivalent to 85% of the one-repetition maximum (1RM) per exercise (high intensity training sessions). The perceived exertion level on the OMNI-RES scale progressed from 6-7 (somewhat hard) in the first 4 weeks to 8-9 (hard) in the remaining 16 weeks. Control of the intensity by this method (which takes into account the grip width, band color, and number of bands) has been previously validated in young adults, middle aged adults, and older adults, and will be the first time that it will be used the validate scale for older adults in the intervention training. The number of sets per exercise progressed from 3 in the first 8 weeks to 4 in the remaining 12 weeks in both groups, with 120s of active recovery (slow rhythmic swinging of the extremities without the use of elastic bands) between sets and 90s of rest between exercises. The speed of execution of the exercises was controlled using a metronome marking the cadence (2s of concentric contraction and 2s of eccentric contraction). The training session will consist in a general warm-up, 6 resistance exercises, including 2 upper limb exercises (elbow curl and chest press), 2 lower limb exercises (lunge and standing hip abduction), and 2 exercises combining both upper and lower limbs at the same time (squat plus upright rowing and squat plus shoulder press) and finally the cooldown routine. Primarily multijoint exercises were chosen to emphasize both major and minor muscle groups.

The H-SPEED group will perform the same routine than the TRADICIONAL group (the same general warm-up, the same 6 resistance exercises and the same cooldown routine) with the difference that this group will perform the concentric phase of each repetition in the resistance exercises ''as fast as possible'', will pause for 1 second, and will perform the eccentric phase in 2-3 seconds (the speed of execution of the exercises was controlled using a metronome). This group will perform 12 submaximal repetitions with very low perceived exertion (3 of 10) and ''rapid´´ in the qualitative perceived exertion scale for power training, equivalent to 40-50% 1RM (low-intensity). The number of sets per exercise progressed from 3 in the first 8 weeks to 4 in the remaining 12 weeks, with 90s of active recovery between sets (slow rhythmic swinging of the extremities without the use of elastic bands) and 60s of rest between exercises.

The MULTICOMPONENT group sessions will include a resistance training component, but will combine it with additional exercise regimens including balance, aerobic, flexibility and coordination. Participants will perform, in this order, balance exercises followed by resistance/coordination, aerobic/coordination and flexibility exercises in each session. The balance training will consist in static, dynamic and proactive balance exercises. In the resistance training block, the participants will perform 15 submaximal repetitions with a perceived exertion level on the OMNI-RES Scale 6-7 (somewhat hard) in the first 8 weeks and 8-9 (hard) in the remaining 12 weeks. Participants will perform 2 resistance exercises (squat plus upright rowing and lunge) at traditional slow-speed (2s of concentric contraction and 2s of eccentric contraction). The number of sets per exercise will progress from 3 in the first 8 weeks to 4 in the remaining 12 weeks, with 90s of active recovery between sets and 60s of rest between exercises. Given the demonstrated importance of reproducing the different challenges encountered in daily life, will be proposed in the aerobic part of the session exercises that will require moving through space using walking progressively at faster speeds to light skipping, jogging, or with longer steps, and while adding the use of the arms. The heart rate will be monitored by the polar team system, which allows monitoring the heart rate of different people at the same time. The intensity of this part will progress from 65 to 85% of the maximum heart rate over the training weeks. The flexibility block will consist in static stretching exercises of upper and lower limbs. Finally, the coordination exercises will be performed in the rests periods of resistance and aerobic blocks, and will consist of psychomotor (reaction time) exercises, dance movements and obstacle exercises. Specific cognitive challenges were integrated also into this block (coordination) to engage executive function, and to specifically stimulate the inhibition of habitual responses and cognitive flexibility. For instance, participants will have to perform task sequences while reversing or ''scattering'' a learned order, or to learn different stimulus-response associations and then switch between them according to external cues. The difficulty of balance and coordination exercises will increase progressively to generate adaptations.

The subjects will perform four sessions of pre-intervention familiarization to (a) select the color, grip width, and number of bands; (b) adapt the rate of perceived exertion; and (c) learn the correct technique for the exercises. The loads will be adjusted every week to maintain the appropriate training intensities by adapting the color and number of elastic bands along with the grip width. Training attendance will be recorded at every session. All the training sessions will be performed in two Municipal Activity Centers for Older People located in Valencia (Campanar and Nou Benicalap centers), under the supervision of a qualified and experienced sports scientist and physiotherapists to ensure safety and compliance.

All the supervised programs will include 2 weekly sessions will perform on nonconsecutive days (separated by 48-72 hr) for 20 weeks. Each session will be performed in groups, and each participant always will perform the exercises in the same order, alternating between the upper and lower limbs. Elastic bands (TheraBand®, Akron, OH, USA) and chairs will be used as the equipment.

ELIGIBILITY:
Inclusion Criteria:

* Age>60 years.
* Physically independent (able to walk 100 meters without a walking aid and climb 10 steps without rest).
* Medical certificate of suitability or fitness to practice resistance training activities.
* No plans to leave the area during the intervention.
* Cognitive ability to understand, follow the instructions and sign the informed consent form.
* Free of any antioxidant supplements for at least 6 weeks before the start of this study.
* Willingness to be randomized to either intervention group and to follow the study protocol.

Exclusion Criteria:

* Presence of cardiovascular, musculoskeletal, renal, liver or neuromuscular disorders that would prevent the participant from performing the exercises.
* Body weight changes >10% in the previous year.
* Intake of prescription medications that were expected to alter the results of the study (ergogenic, dietary aids, estrogen, steroid hormones, calcitonin, or corticosteroids).
* A history of malignant neoplasms.
* Engagement in regular strength training (more than once a week) during the previous 6 months.
* Individuals participating in another research project (within the last 6 months) involving dietary, exercise and/or pharmaceutical intervention
* Mini Mental State Examination lower than 24/30
* Severe visual or hearing impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in DNA oxidative stress | Baseline and 20 weeks
  The oxidative stress of DNA will be assessed via urine collections of 8-oxo-7,8- dihydro-20-deoxyguanosine (8-OHdG) in nmol/mmol creatinine.
Change in lipid peroxidation | Baseline and 20 weeks
  The lipid peroxidation will be assessed via urine and blood collections of 8-isoprostane(nmol /mmol creatinine) and Malondialdehyde (μmol/L)
Change in protein oxidation | Baseline and 20 weeks
  The protein oxidation will be assessed via blood collections of protein carbonyl (nmol/L)
Change in antioxidants enzymes | Baseline and 20 weeks
  The antioxidants enzymes will be assessed via blood collections of superoxid dismutase (U · mL-1), reduced glutathione (nmol/mg protein), glutathione peroxidase (IU/g Hb), oxidized glutathione (nmol/mg protein), and catalase (IU/g Hb).
Change in metabolic profile | Baseline and 20 weeks
  The metabolic profile will be assessed via blood collections of glycosylated hemoglobin A1C (%) and basal glucose (mmol/l).
Change in lipid profile | Baseline and 20 weeks
  The lipid profile will be assessed via blood collections total cholesterol (mg/dL), high-density lipoprotein cholesterol (mg/dL), low-density lipoprotein cholesterol (mg/dL) and triglycerides (mg/dL).
Change in immune profile | Baseline and 20 weeks
  The immune profile will be assessed via blood collections of platelet counts (10*9/L), plateletcrit (%), mean platelet volum (fl), platelet distribution width (%), leukocytes (% and 10*9/L), neutrophils (% and 10*9/L), lymphocytes (% and 10*9/L), monocytes (% and 10*9/L), eosinophils (% and 10*9/L), basophils (% and 10*9/L).
Change in C-reactive Protein | Baseline and 20 weeks
  The C-reactive protein (mg/L) will be assessed via blood collections.
Change in bone metabolism | Baseline and 20 weeks
  The bone metabolism will be assessed via blood collections of osteocalcine, and beta crosslaps.
Change in muscle strength | Baseline and 20 weeks
  The dynamic maximal concentric muscle strength of the dominant side of hip (abduction and adduction muscle groups), knee and elbow (flexion and extension muscle groups) will be measured with an isokinetic dynamometer (Biodex System 4 Pro; Biodex, Shirley, NY) at two angular velocities, 60°/s and 180°/s. Maximal voluntary concentric isokinetic torque will be assessed in Newton-meters (N-m). The isometric maximal muscle hand grip strength of both hands will be measured with a dynamometer.
Change in functional performance | Baseline and 20 weeks
  The functional performance will be assessed with Senior Fitness tests that involve 6 tests: Arm Curl (number of biceps curl in 30 seconds); Chair Stand (stand up from a chair as often as possible within 30s); Back Scratch (for shoulder flexibility, cm between fingertips in the back); Chair sit and reach (for lower flexibility, cm between the extended middle fingers and the tip of the shoe); Up-and-Go (for dynamic balance, time for got up from the chair, walk as quickly as possible around a cone placed 2.4 m from the chair, and resume the seated position); Six-Minute walking test (for aerobic capacity, distance walked in 6 minutes).
Change in lower extremity performance | Baseline and 20 weeks
  The lower extremity performance will be assessed with the Short Physical performance battery (SPPB). The SPPB includes an assessment of standing balance, a timed 2.4-meter walk, and a timed test of 5 repetitions of rising from a chair and sitting down (chair-5 time). Each of the three tests is scored, based on performance between 0 and 4, leaving a maximum score of 12 for those individuals performing at the highest levels. Times, measured to the nearest 0.1 second using a stopwatch, for the 2.4-meter walk and chair stand will be used to calculate gait speed and chair-5 time. Balance will be assessed using unilateral stance where subjects are instructed to stand unsupported on the leg of their choice. Time that the leg is off the ground will be recorded.

SECONDARY OUTCOMES:
Change in 10-meters walking speed | Baseline and 20 weeks
  The 10-meters walking speed will be assessed outdoors over a course of 10 m and the time will be recorded. Habitual and maximal walking speeds will be assessed two times by asking participants to walk respectively at ''the speed at which you would walk to the shops'' and ''as fast as possible without running''.
Change in stair climbing | Baseline and 20 weeks
  The time to walk up one flight of stairs will be measured by having the participants walk up one flight of stairs consisting of 23 steps as quickly as possible. The time to complete this task will be recorded to the nearest hundredth of a second using a handheld stopwatch.
Change in muscle thickness | Baseline and 20 weeks
  Muscle thickness (cm) of rectus femoris and biceps brachii of the of the dominant side will be assessed by B-Mode ultrasound (E-Cube 7, Alpinion Medical Systems Co, Seoul, Korea)
Change in pennation angle | Baseline and 20 weeks
  Pennation angle (°) of rectus femoris and biceps brachii of the of the dominant side will be assessed by B-Mode ultrasound (E-Cube 7, Alpinion Medical Systems Co, Seoul, Korea).
Change in cross-sectional area | Baseline and 20 weeks
  Cross-sectional area (cm2) of rectus femoris and biceps brachii of the of the dominant side will be assessed by B-Mode ultrasound (E-Cube 7, Alpinion Medical Systems Co, Seoul, Korea)
Change in fascicle length | Baseline and 20 weeks
  Fascicle length (cm) of rectus femoris and biceps brachii of the of the dominant side will be assessed by B-Mode ultrasound (E-Cube 7, Alpinion Medical Systems Co, Seoul, Korea)
Change in echo intensity | Baseline and 20 weeks
  Echo intensity of rectus femoris and biceps brachii of the of the dominant side will be assessed by B-Mode ultrasound (E-Cube 7, Alpinion Medical Systems Co, Seoul, Korea). Echo Intensity of the rectus femoris and vastus lateralis will be obtained using the same images as for cross-sectional area. Echo intensity will be determined by grayscale analysis using the standard histogram function in ImageJ. Echo intensity in the region of interest will be expressed as arbitrary unit values between 0-255 (0: black; 255: white).
Change in total mass | Baseline and 20 weeks
  Total mass (Kg) will be assessed for whole body and appendicular regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in fat mass | Baseline and 20 weeks
  Fat mass (Kg) will be assessed for whole body and appendicular regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in fat free mass | Baseline and 20 weeks
  Fat free mass (Kg) will be assessed for whole body and appendicular regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in percentage of fat mass | Baseline and 20 weeks
  Percentage of fat mass will be assessed for whole body and appendicular regions using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in waist circumference | Baseline and 20 weeks
  Waist circumference will be measured at the midpoint between the lower margin of the least palpable rib and the top of the iliac crest, using a stretch-resistant tape that provides a constant 100g tension in cm.
Change in hip circumference | Baseline and 20 weeks
  Hip circumference will be measured around the widest portion of the buttocks, with the tape parallel to the floor, using a stretch-resistant tape that provides a constant 100 g tension in cm.
Change in waist/hip ratio | Baseline and 20 weeks
  Waist/hip ratio will be assessed by dividing waist circumference by hip circumference.
Change in waist/height ratio | Baseline and 20 weeks
  Waist/height ratio will be assessed by dividing waist circumference by height.
Change in weight | Baseline and 20 weeks
  Weight will be recorded to the nearest 0.01 Kg, using a Tanita® BC-418MA digital scale (Tanita Corp., Tokyo, Japan).
Height | Baseline
  Height will be recorded to the nearest 0.01 cm using a stadiometer (Seca 711, Hamburg, Germany)
Change in body mass index (BMI) | Baseline and 20 weeks
  BMI will be calculated as body weight (kilogram) divided by height (meter) squared (kilogram per square meter).
Change in bone mineral density (BMD) | Baseline and 20 weeks
  BMD (g/cm2) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Ward's triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change bone mineral content (BMC) | Baseline and 20 weeks
  BMC(g) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Ward's triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change T-Score | Baseline and 20 weeks
  T-Score (SD) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Ward's triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in Z-Score | Baseline and 20 weeks
  Z-Score (SD) will be assessed for whole body, proximal femur on the non-dominant side (femoral nech, trochanter, intertrochanter, Ward's triangle and total hip) and lumbar spine segments (L1-L4) (L2-L4) (L1-L3) and single vertebrae (L1, L2, L3, L4) will be assessed using a dual-energy-X ray fan beam absorptiometry (QDR® Hologic Discovery Wi, Hologic Inc., Waltham, MA, USA) equipped with APEX software (APEX Corp., version 12.4, Waltham, MA, USA).
Change in fracture risk | Baseline and 20 weeks
  Will be assessed via the FRAX ® tool.
Change in static balance | Baseline and 20 weeks
  Static steady-state balance will be assessed with One-legged stance (OLST) and the Sharpened Romberg test. The OLST will be performed in the standing position, and start when the subjects lift the appropriate foot off the ground. Timing will stop if the subjects displace the foot they will be standing on, touch the suspended foot to the ground, use the suspended foot to support the weight-bearing limb, or reached the maximum balance time of 30 seconds. The participants will perform each test with their eyes open and closed, and both will be performed with the shoes-on and shoes-off conditions. For the Sharpened Romberg test participants will stand erect on a level surface wearing flat shoes with his or her feet aligned in a strict tandem heelto-toe position, arms crossed over the chest, and the open palm of the hand falling on the opposite shoulder. Once stable, the subject will close his or her eyes and will try to maintain that position for 60 seconds.
Self-reported falls | Baseline and 20 weeks
  Self-reported falls will be assessed by the total number of falls during the study period.
Rate of falls | Baseline and 20 weeks
  Rate of falls will be assessed by the total number of falls during the training period compared to the number of falls during the year before the participation on the study.
Self-perceptions of physical activity | At week 20
  Self-perceptions of the physical activity (training mode) will be assessed by a questionnaire designed by the researchers of the project.
Change in self-reported quality of life | Baseline and 20 weeks
  Will be assessed via Short form quality of life questionnaire (SF36)
Change in self-reported sleep quality | Baseline and 20 weeks
  Will be assessed via The Pittsburgh Sleep Quality Index, a self-rated sleep questionnaire for measuring sleep quality.
Change in self-reported anxiety | Baseline and 20 weeks
  Will be assessed via Overall Anxiety Severity and Impairment Scale (OASIS), a five-item self-report measure of anxiety severity and resulting functional impairment. Scores on the measure range from 0 to 20, with higher scores indicating greater anxiety-related severity and impairment.
Change in self-reported depression | Baseline and 20 weeks
  Will be assessed via Overall Depression Severity and Impairment Scale (ODSIS). The ODSIS was developed to assess depression in the following domains: frequency (Item 1), intensity (Item 2), functional impairment in pleasurable activity (Item 3), work or school (Item 4), and interpersonal relationships (Item 5). Items of ODSIS are scored on a five-point Likert scale of 0-4. Scores on the measure range from 0 to 20, with higher scores indicating greater depression-related severity and impairment.
Change in basic activities of daily living | Baseline and 20 weeks
  Will be assessed via Barthel index of activities of daily living.
Change in instrumental activities of daily living | Baseline and 20 weeks
  Will be assessed via Lawton and Brody instrumental activities of daily living scale. There are eight domains of function measured with the Lawton and Brody scale. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent).
Nutritional assessment | Baseline and 10 weeks
  Nutritional status will be assessed by a 3-day diet records over 2 weekdays and 1 weekend day. Diet records will be analyzed using the program DIAL 3.5.0.3 (ALCE INGENIERIA, Madrid, Spain).
Adherence to the Mediterranean diet | Baseline and 10 weeks
  Adherence to the Mediterranean diet will be assessed by PREDIMED adherence to the Mediterranean diet questionnaire.

OTHER OUTCOMES:
Level of physical activity | Baseline
  The level of physical activity of the participants will be assessed by Global Physical Activity Questionnaire (GPAQ)
Cognitive function | Baseline
  The cognitive function will be assessed by the Mini Mental State Examination (MMSE) questionnaire.
Attendance to training sessions | From week 1 to week 20
  Daily training session attendance records will be collected by the instructors.
Adherence to training program | At week 20
  Adherence levels will be calculated at the end of the training period. Nonadherence is define as "those not attending at follow-up and have not attend for 4 weeks during the training period, and have not given a reason for nonattendance or those who have stated they are dropping out."
Heart rate during the training exercise sessions | From week 1 to week 20
  The heart rate will be monitored by the Polar Team System, which allows monitoring the heart rate of different people at the same time.
Rating of perceived exertion | From week 1 to week 20
  Will be assessed the perceived exertion during the training sessions asking the level of perceived on the OMNI-RES Scale validated for older adults.
Change in number of medication used | Baseline and 20 weeks
  Will be recorded the number of medication used for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Colado Sánchez, Full professor, Principal Investigator — University of Valencia
Locations (3):
- Spain (3):
  - Faculty of Physical Activity and Sports Sciences, Valencia
  - Municipal Center of Activities for Older People of Campanar, Valencia
  - Municipal Center of Activities for Older People of Nou Benicalap, Valencia

REFERENCES:
- [Derived] Gargallo P, Tamayo E, Jimenez-Martinez P, Juesas A, Casana J, Benitez-Martinez JC, Gene-Morales J, Fernandez-Garrido J, Saez GT, Colado JC. Multicomponent and power training with elastic bands improve metabolic and inflammatory parameters, body composition and anthropometry, and physical function in older women with metabolic syndrome: A 20-week randomized, controlled trial. Exp Gerontol. 2024 Jan;185:112340. doi: 10.1016/j.exger.2023.112340. Epub 2023 Dec 11. PMID 38061437